CLINICAL TRIAL: NCT02644499
Title: Comparison of Combination Disease Modifying Antirheumatic Drugs (DMARDs) With Single Drug (Methotrexate) Therapy in Early Rheumatoid Arthritis
Brief Title: Comparison of Combination Disease Modifying Antirheumatic Drugs With Methotrexate Therapy in Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr. Vir Singh Negi, Professor and head of the department, Department of Clinical Immunology, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIP/IEC/SC/2013/5/433
Record Dates: First submitted 2015-12-30; First posted 2015-12-31 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Leflunomide; Hydroxychloroquine; Prednisolone; Steroids; Glucocorticoids; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination therapy (Active Comparator): Combination of Methotrexate (up to 25 mg per week), Leflunomide (20 mg once a day) and Hydroxychloroquine (200-400 mg once at night). All drugs are to be taken orally. Duration of therapy is for 3 months. All patients will receive folic acid (5 mg twice a week) along with methotrexate. Low dose prednisolone (weeks 1-2: 15 mg/day, weeks 2-4: 10 mg/day, weeks 4-6: 5 mg/day and weeks 6-8: 2.5 mg/day then stop) will be given as bridging therapy.
  Interventions: Drug: Methotrexate; Drug: Leflunomide; Drug: Hydroxychloroquine; Drug: Prednisolone; Drug: Folic Acid
- Monotherapy (Active Comparator): Methotrexate (up to 25 mg once a week) for 3 months. All patients will receive folic acid (5 mg twice a week) along with methotrexate. Low dose prednisolone (weeks 1-2: 15 mg/day, weeks 2-4: 10 mg/day, weeks 4-6: 5 mg/day and weeks 6-8: 2.5 mg/day then stop) will be given as bridging therapy.
  Interventions: Drug: Methotrexate; Drug: Prednisolone; Drug: Folic Acid

INTERVENTIONS:
Drug: Methotrexate — Methotrexate, a structural analogue of folic acid, can be administered orally or parenterally to treat a variety of rheumatic dise
  Other Names: Folitrax, MTX
Drug: Leflunomide — Leflunomide inhibits pyrimidine synthesis, resulting in blockade of T-cell proliferation. Leflunomide is used in patients with moderate to severe active rheumatoid arthritis with early or late disease
  Other Names: Arava, Lefno
  Arms: Combination therapy
Drug: Hydroxychloroquine — Hydroxychloroquine (HCQ) is a well-tolerated DMARD that is commonly used in combination therapy regimens for RA. HCQ is more commonly used than chloroquine.
  Other Names: HCQ
  Arms: Combination therapy
Drug: Prednisolone — Low dose prednisolone (weeks 1-2: 15 mg/day, weeks 2-4: 10 mg/day, weeks 4-6: 5 mg/day and weeks 6-8: 2.5 mg/day then stop)
  Other Names: Steroids, Glucocorticoids
Drug: Folic Acid — Folic acid is to be given to all patients receiving methotrexate at a dose of 5 mg twice a week.
  Other Names: Folvite, Folate

SUMMARY:
This study will be conducted to find out how well a patient of rheumatoid arthritis (RA) will respond to disease-modifying antirheumatic drugs (DMARDs). RA is a chronic inflammatory arthritis, which leads to joint damage & disability if not treated properly. A DMARD is used to treat RA that slows down or prevents joint damage, as opposed to just relieve pain or inflammation by painkillers. The study will be conducted at the Department of Clinical Immunology, JIPMER (Jawaharlal Institute of Postgraduate Medical Education & Research). Patients will receive either a single DMARD (Methotrexate) or combination DMARDs therapy (Methotrexate + Leflunomide + Hydroxychloroquine). During treatment course, routine blood investigations will be carried out to monitor treatment response and side effects.

DETAILED DESCRIPTION:
Patients aged ≥18 years, fulfilling the 2010 ACR EULAR criteria for RA (symptom duration less than one year) & having moderate to severe disease activity (DAS28≥3.2) will be invited to participate. After providing written informed consent, eligible patients will be stratified into two groups. Block randomization will be done to generate random allocation sequence.

Treatment Group I will be treated with Methotrexate (MTX) monotherapy and Treatment Group II will be treated with Methotrexate + Leflunomide (LEF) + Hydroxychloroquine (HCQ) combination therapy. Concurrent treatment with non-steroidal anti-inflammatory drugs in adequate dose and oral low dose Glucocorticoids (GC) (max: 15 mg/d) will be allowed during the study.

DMARD dosages used are: MTX 25 mg/week orally (dosage after 6 weeks), LEF 20 mg/day (dosage after 2 weeks) and HCQ 400 mg/day. GCs will be given in an oral tapering scheme. All patients will be prescribed folic acid (10 mg/week) during MTX prescription.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years satisfying 2010 ACR (American college of rheumatology) - EULAR criteria for RA
2. Arthritis in one or more joint (s)
3. Symptom duration <1 year
4. DMARD naive
5. Patients with moderate to severe disease activity (DAS28 ≥3.2)

Exclusion Criteria:

1. Disease in Remission/inactive disease (DAS28 criteria)
2. End stage disease (deformed fixed joints)
3. Patients with vasculitis or other severe extra-articular features
4. Contraindications to DMARD therapy (Chronic Alcoholism, Chronic liver disease, Evidence of acute/chronic infection, Chronic kidney disease, Patients with leucopenia (<3.0×109/l), thrombocytopenia (<150×109/l), aspartate aminotransferase (AST)/alanine aminotransferase (ALT)>2× upper normal value and creatinine level >150 μmol/l )
5. Pregnant, lactating females or inadequate contraception
6. Patients unable to come for regular follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
A good response according to European league against rheumatism (EULAR) response criteria and Functional ability with Indian health assessment questionnaire (iHAQ) | 3 months
  A good response is defined as a decrease after randomization of disease activity score- 28 joints (DAS28) score by >1.2, and a resulting DAS28 score ≤ 3.2.
  Indian version of HAQ (iHAQ) has been validated in patients with RA, which comprises 12 questions (nine basic and three advanced activity of daily living) relevant to the Indian population. For each question there is a four-level difficulty scale ranging from 0 to 3 that represent no difficulty ('0'), some difficulty ('1'), much difficulty ('2'), and inability to do ('3'). The final score is the mean of the highest scores across the eight categories and ranges from 0 to 3, with higher levels indicating more disability.

SECONDARY OUTCOMES:
Mean changes over time in early morning stiffness (EMS) | 3 months
Mean changes over time in erythrocyte sedimentation rate (ESR) | 3 months
Disease activity as per ultrasound (US-7) score | 3 months
Radiographic progression assessed with Simple Erosion Narrowing Score (SENS) | 3 months
Adverse drug reactions | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vir S Negi, DM, Principal Investigator — Jawaharlal Institute of Postgraduate Medical Education & Research; Jignesh B Usdadiya, MD, Study Chair — Jawaharlal Institute of Postgraduate Medical Education & Research
Locations (1):
- Jawaharlal Institute of Postgraduate Medical Education & Research (JIPMER), Puducherry, Pondicherry UT, India

IPD SHARING:
Plan to Share IPD: No